CLINICAL TRIAL: NCT06852352
Title: A Prospective, Single-center, Single-arm, Exploratory, 24-Month Study to Confirm Efficacy of Modified Deep Cervical Lymphovenous Anastomosis (LVA) in Subjects with Alzheimer's Disease/ Parkinson's Disease
Brief Title: An Exploratory Study to Confirm Efficacy of Modified Deep Cervical Lymphovenous Anastomosis (LVA) in Alzheimer's Disease/ Parkinson's Disease
Acronym: SOLVEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Zybio Inc. (Unknown)
Responsible Party: Principal Investigator, Youmao Zheng, MM, Head of Lymphatic and Microsurgical Reconstructive Surgery, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2025008
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Parkinson Disease
Keywords: LVA
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The clinically diagnosed patients with MCI or mild-moderate dementia caused by AD/PD (Experimental)
  Interventions: Procedure: Modified deep cervical Lymphatic-Venous Anastomosis

INTERVENTIONS:
Procedure: Modified deep cervical Lymphatic-Venous Anastomosis — Deep cervical lymph-vein anastomosis surgery, connecting deep cervical lymph input vein vessels to enhance glymphatic-mediated protein clearance

SUMMARY:
Alzheimer's disease (AD) and Parkinson's disease (PD) are characterized by pathological protein accumulation in the brain-Aβ/tau in AD and α-synuclein in PD. Recent studies have indicated that age-related lymphatic vessel atrophy compromises the metabolic clearance capacity of meningeal lymphatic vessels, potentially disrupting the equilibrium between production and clearance of Aβ/α-synuclein, ultimately leading to pathological accumulation of these proteins within the brain. Deep cervical lymphovenous anastomosis (LVA), a surgical technique proven effective in restoring lymphatic drainage in lymphedema, may enhance clearance of neurotoxic proteins by improving cervical lymphatic outflow. This project aims to evaluate the efficacy of modified deep cervical LVA in treating AD and PD, establishing a novel therapeutic strategy to modify disease progression and improve quality of life in neurodegenerative disorders, additionally offering the pathogenic mechanisms underlying neurodegenerative disorders.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) and Parkinson's disease (PD) are progressive neurodegenerative disorders characterized by pathological protein aggregation-Aβ plaques and tau tangles in AD, and α-synuclein Lewy bodies in PD. Emerging evidence implicates that the glymphatic-meningeal lymphatic system and deep cervical lymph nodes constitute the central pathway for metabolite clearance of cerebral macromolecules. Aging-associated lymphatic vessel atrophy disrupts the equilibrium between protein production and clearance, exacerbating neurotoxicity. Deep cervical lymphovenous anastomosis (LVA), a surgical technique validated in lymphedema management, aims to restore cervical lymphatic drainage and enhance glymphatic-mediated protein clearance. This study investigates the therapeutic potential of modified deep cervical LVA in AD and PD. A prospective cohort will undergo modified deep cervical LVA with longitudinal assessments, including cerebrospinal fluid (CSF) and plasma biomarkers (Aβ42, p-tau181, p-tau217, GFAP, NfL, α-synuclein), neuroimaging (MRI and PET-CT), and clinical endpoints (CDR, MMSE, MoCA, BADL and IADL for AD, UPDRS and PDQ-39 for PD). Mechanistically, we hypothesize that modified deep cervical LVA will reduce intracranial pressure gradients, augment meningeal lymph flow, and accelerate interstitial waste drainage, thereby mitigating neuroinflammation and neuronal damage. This trial aims to verify the efficacy of modified deep cervical LVA to modify disease progression in AD and PD, providing a surgically scalable approach to delay progression of neurodegenerative disorders and improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

Alzheimer's disease:

1. Male or female, the age ranged from 50 to 75 years old
2. Informed consent signed and dated by patient or legal representative
3. Patients diagnosed principally with mild cognitive impairment or dementia caused by Alzheimer's disease
4. Positive result of Amyloid PET imaging (Centiloids ≥37)
5. HAMD score ≤17
6. Hachinski score ≤4 Patients who meet ASA (American Society of Anesthesiologists) grade I-III criteria

Parkinson's disease:

1. Male or female, the age ranged from 50 to 80 years old
2. Informed consent signed and dated by patient or legal representative
3. Patients diagnosed with Parkinson's disease or probable Parkinson's disease according to the Clinical Diagnostic Criteria for Parkinson's Disease in China (2016) or MDS
4. Stage I-IV patients according to Hoehn and Yahr Scale
5. Patients documented history of Parkinson's disease for more than 2-5 years to ensure clinical stability of symptoms and exclude the possibility of early misdiagnosis of other conditions

Exclusion Criteria:

1. Contraindications for MRI, ICG angiography, or PET scanning
2. Contraindications for lumbar puncture
3. Functional impairment of vital organs (cardiac, pulmonary, renal, hepatic), including reduced left ventricular ejection fraction, prolonged QT interval, severe pulmonary diseases, and severe hepatic/renal insufficiency
4. MRI results suggesting intracranial active/acute pathologies, including infections, space-occupying lesions, major hemorrhages, or ≥4 lobar microhemorrhages;
5. Conditions predisposing to increased intracranial hemorrhage risk, such as hematological disorders, hemorrhagic/coagulation disorders;
6. Poorly controlled thyroid dysfunction;
7. Cerebrovascular or systemic vasculopathy;
8. Severe cardiac disease or hemodynamic instability;
9. Uncontrolled severe hypertension;
10. Substance use disorders (including illicit drugs, anesthetics, and alcohol dependence);
11. Active severe infections, including HIV positivity and acute critical infections;
12. Severe psychiatric disorders or significant suicide risk;
13. Chronic hypnotic use (more than twice weekly for over one month);
14. History of untreated/uncured malignancies;
15. Participation in other interventional clinical trials within preceding 3 months;
16. Poor compliance with inability/unwillingness to complete scheduled postoperative follow-ups;
17. Other investigator-determined contraindications for trial participation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's disease: Change in Clinical Dementia Rating Scale sum of the boxes (CDR-SB) | up to 2 years
  The Clinical Dementia Rating Scale sum of the boxes (CDR-SB) will be used to evaluate the general cognitive function. CDR-SB ranges from 0 to 18, and higher value represents a worse outcome.
Alzheimer's disease: Change in Mini-mental State Examination (MMSE) | up to 2 years
  The Mini-mental State Examination (MMSE) will be used to evaluate the general cognitive function. MMSE ranges from 0 to 30, and higher value represents a better outcome.
Alzheimer's disease: Change in Montreal Cognitive Assessment (MoCA) | up to 2 years
  The Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.
Alzheimer's disease: Change in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (Severe Version) (ADCS-ADL-SEV) | up to 2 years
  The ADCS-ADL-SEV consists of 19 items. Ratings reflect caregiver observations about the patient's actual functioning over the previous month and provide an assessment of change in the functional state of the participant over time. The total score ranges from 0 to 54, with lower values over time reflecting functional deterioration.
Parkinson's disease：Change in Unified Parkinson's Disease Rating Scale (UPDRS) | up to 2 years
  The scale assesses the functional status of patients with parksinon´s disease, including the independency of daily activities, mood, secondary effects of medications and motor complications. The total UPDRS score ranges from 0 to 199 points, with higher scores indicating more severe symptoms.
Parkinson's disease：Change in The Hoehn and Yahr Scale | up to 2 years
  The Hoehn and Yahr (H&Y) scale is the most widely used and universally accepted staging system for overall functional disability in Parkinson's disease. The H&Y Scale categorizes Parkinson's disease progression into 7 stages. Each stage reflects worsening motor function and loss of independence.
Parkinson's disease：Change in Parkinson's Disease Questionnaire-39 (PDQ-39) | up to 2 years
  The Parkinson's Disease Questionnaire-39 (PDQ-39) is a vital tool for assessing the quality of life in Parkinson's disease patients. The total score ranges from 0 to 100 points, with higher scores indicating worse quality of life.

SECONDARY OUTCOMES:
Alzheimer's disease: Change in amyloid deposit in brain | baseline, 1year, 2 years
  Change from baseline as measured by amyloid positron emission tomography (PET) scan using centiloids. The centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan. A negative change indicates an improvement from baseline.
Alzheimer's disease: Change in brain Tau deposition in a subset of participants | baseline, 1year, 2 years
  Change from baseline as measured by Tau PET scan
Alzheimer's disease: Change in fluid biomarker | up to 2 years
  Change from baseline in cerebrospinal fluid (CSF)/plasma p-tau217, p-tau181, Aβ42, GFAP and NfL levels
Alzheimer's disease: Change in Neuropsychiatric Inventory (NPI-Q) Total Severity Score | up to 2 years
  The NPI-Q is a brief, caregiver-reported assessment of neuropsychiatric symptoms associated with dementia. The NPI-Q yields total scores for Severity and Distress, reflecting the sum of ratings across all domains, with higher scores indicating a greater degree of symptom severity and caregiver distress, respectively.
Alzheimer's disease: Change in Clinical Global Impression | up to 2 years
  The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) is used to assess the severity and progression of AD, where scores from 0 to 7 represent the spectrum of symptom intensity (0 = asymptomatic to 7 = extremely severe). The Efficacy Index (EI), a composite metric balancing therapeutic benefits and side effects, ultimately reflects the efficacy of surgical interventions for AD.
Alzheimer's disease: Changes in the functional connectivity in brain in a subset of participants | baseline, 1year, 2 years
  Change from baseline in disrupted functional connectivity as measured by functional MRI (fMRI)
Parkinson's disease: Change in fluid biomarker | up to 2 years
  Change from baseline in cerebrospinal fluid (CSF)/plasma α-synuclein, GFAP, NfL levels
Changes in the hippocampal volume | baseline, 1year, 2 years
  Change from baseline in hippocampal volume (mm3) as measured by structural Magnetic Resonance Imaging (sMRI)
Changes in the cortical thickness | baseline, 1year, 2 years
  Change from baseline in cortical thickness (mm) as measured by structural Magnetic Resonance Imaging (sMRI)
Changes in the water diffusion characteristics in brain | baseline, 1year, 2 years
  Change from baseline in water diffusion reflects the White Matter Hyperintensities (WMH)/efficiency of lymphatic drainage as measured by MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Li Y, Wang L, Zhong J, Xu H, Han Y; Alzheimer's Disease Neuroimaging Initiative; Zuo C, Jiang J. Impaired glymphatic function as a biomarker for subjective cognitive decline: An exploratory dual cohort study. Alzheimers Dement. 2024 Sep;20(9):6542-6555. doi: 10.1002/alz.14149. Epub 2024 Aug 6. PMID 39107995
- [Background] Huang SY, Zhang YR, Guo Y, Du J, Ren P, Wu BS, Feng JF; Alzheimer's Disease Neuroimaging Initiative; Cheng W, Yu JT. Glymphatic system dysfunction predicts amyloid deposition, neurodegeneration, and clinical progression in Alzheimer's disease. Alzheimers Dement. 2024 May;20(5):3251-3269. doi: 10.1002/alz.13789. Epub 2024 Mar 19. PMID 38501315
- [Background] Pappolla M, Sambamurti K, Vidal R, Pacheco-Quinto J, Poeggeler B, Matsubara E. Evidence for lymphatic Abeta clearance in Alzheimer's transgenic mice. Neurobiol Dis. 2014 Nov;71:215-9. doi: 10.1016/j.nbd.2014.07.012. Epub 2014 Aug 4. PMID 25102344
- [Background] Nedergaard M, Goldman SA. Glymphatic failure as a final common pathway to dementia. Science. 2020 Oct 2;370(6512):50-56. doi: 10.1126/science.abb8739. PMID 33004510
- [Background] Iliff JJ, Wang M, Liao Y, Plogg BA, Peng W, Gundersen GA, Benveniste H, Vates GE, Deane R, Goldman SA, Nagelhus EA, Nedergaard M. A paravascular pathway facilitates CSF flow through the brain parenchyma and the clearance of interstitial solutes, including amyloid beta. Sci Transl Med. 2012 Aug 15;4(147):147ra111. doi: 10.1126/scitranslmed.3003748. PMID 22896675
- [Background] Aspelund A, Antila S, Proulx ST, Karlsen TV, Karaman S, Detmar M, Wiig H, Alitalo K. A dural lymphatic vascular system that drains brain interstitial fluid and macromolecules. J Exp Med. 2015 Jun 29;212(7):991-9. doi: 10.1084/jem.20142290. Epub 2015 Jun 15. PMID 26077718
- [Background] Chen F, Xie X, Wang L. Research Progress on Intracranial Lymphatic Circulation and Its Involvement in Disorders. Front Neurol. 2022 Mar 14;13:865714. doi: 10.3389/fneur.2022.865714. eCollection 2022. PMID 35359624
- [Background] Zhao H, Sun M, Zhang Y, Kong W, Fan L, Wang K, Xu Q, Chen B, Dong J, Shi Y, Wang Z, Wang S, Zhuang X, Li Q, Lin F, Yao X, Zhang W, Kong C, Zhang R, Feng D, Zhao X. Connecting the Dots: The Cerebral Lymphatic System as a Bridge Between the Central Nervous System and Peripheral System in Health and Disease. Aging Dis. 2024 Feb 1;15(1):115-152. doi: 10.14336/AD.2023.0516. PMID 37307828
- [Background] Vera Quesada CL, Rao SB, Torp R, Eide PK. Immunohistochemical visualization of lymphatic vessels in human dura mater: methodological perspectives. Fluids Barriers CNS. 2023 Mar 28;20(1):23. doi: 10.1186/s12987-023-00426-3. PMID 36978127
- [Background] Louveau A, Smirnov I, Keyes TJ, Eccles JD, Rouhani SJ, Peske JD, Derecki NC, Castle D, Mandell JW, Lee KS, Harris TH, Kipnis J. Structural and functional features of central nervous system lymphatic vessels. Nature. 2015 Jul 16;523(7560):337-41. doi: 10.1038/nature14432. Epub 2015 Jun 1. PMID 26030524
- [Background] Da Mesquita S, Louveau A, Vaccari A, Smirnov I, Cornelison RC, Kingsmore KM, Contarino C, Onengut-Gumuscu S, Farber E, Raper D, Viar KE, Powell RD, Baker W, Dabhi N, Bai R, Cao R, Hu S, Rich SS, Munson JM, Lopes MB, Overall CC, Acton ST, Kipnis J. Functional aspects of meningeal lymphatics in ageing and Alzheimer's disease. Nature. 2018 Aug;560(7717):185-191. doi: 10.1038/s41586-018-0368-8. Epub 2018 Jul 25. PMID 30046111